CLINICAL TRIAL: NCT05291039
Title: Assessment of Trough Levels and Efficacy of Infliximab and Adalimumab in Inflammatory Bowel Disease Patients.
Brief Title: Infliximab and Adalimumab in Inflammatory Bowel Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Principal Investigator, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Infliximab & Adalimumab in IBD
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Infliximab; Adalimumab
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Intervention Model Description: prospective study for IBD patients receiving either adalimumab (group 1) or infliximab (group 2).
Masking Description: Randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infliximab. (Active Comparator): group 1 (n=20): patients will receive IFX,
  Interventions: Drug: Infliximab
- Adalimumab. (Active Comparator): group 2 (n=20): patients will receive ADA
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Infliximab — group 1 (n=20): patients will receive IFX
  Other Names: IFX
  Arms: Infliximab.
Drug: Adalimumab — group 2 (n=20): patients will receive ADA
  Other Names: ADA
  Arms: Adalimumab.

SUMMARY:
This study aims to assess trough, TREM-1 levels and efficacy of IFX and ADA in IBD patients.

DETAILED DESCRIPTION:
1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University 2. All participants agree to take part in this clinical study, will agree to provide an informed written consent 3. Patients will be divided into 2 treatment groups [group 1 (n=20): patients will receive IFX], [group 2 (n=20): patients will receive ADA]. 4. Statistical tests appropriate to the study will be conducted to evaluate significance of results 5. Results, conclusion, discussion and recommendations will be given

* Type of Study: prospective study for IBD patients receiving either adalimumab or infliximab.
* Study Setting: The Inflammatory Bowel disease outpatient clinic, Tropical Medicine department, Ain Shams University Hospitals.
* Sample Size: Study will be conducted on 40 patients with Inflammatory Bowel Disease (IBD).
* Study procedure

  1. Laboratory investigations

     a) At baseline, all patients will be subjected to i. full history taking regarding: Loss of appetite, abdominal pain, number of motions, bleeding per rectum, number of attacks per year, need for hospitalization per year, Loss of weight, extra intestinal manifestations, anemic manifestations, drug history, ii. Testing the viral markers (HCV Ab, HBs Ag, HB core IgG, HIV) and Tuberculine test or Quantifferon test. (To Exclude latent TB) b) At Baseline and in follow ups, patient will be assessed for the following laboratory investigations: i. Complete blood count (CBC). ii. Liver profile (albumin, INR, total & direct bilirubin, AST, ALT) iii. Kidney function tests e.g BUN and creatinine. iv. Inflammatory Markers (C-reactive protein (CRP), estimated sedimentation Ratio (ESR)).

     v. Stool analysis (WBC's, RBC's, Parasite) vi. Stool culture and sensitivity. vii. Urine analysis. c) Trough concentration of ADA and IFX will be assessed after reaching steady state levels.

     d) TREM-1 levels will be measured for all patients.
  2. Endoscopic intervention

     1. Colonoscopy with terminal ileoscopy with assessment according to Mayo score (loss of vascular pattern, presence of polyps, opacity of mucosa, bleeding on touch, excess exudates, diffuse ulceration, masses, pseudo polyps, site of involvement, linear ulcers, cobblestone appearance, conclusion)
     2. Histopathological examination: (aggregates of PMN's, cryptitis, infiltration of lamina propria, granuloma, depletion of goblet cells, thickened muscularis mucosa, dysplasia & it's degree, malignancy)

Efficacy and safety Assessments

* Target response will be measured according to mucosal healing, ESR and CRP then patients will be reassessed by ECCO guidelines.
* Safety of drugs will be assessed by the monthly follow up of CBC, Liver functions and kidney functions.
* Patients will be asked for the occurrence of any sides in the monthly follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between 18 years and 80 years.
2. Patients having moderate to severe IBD according to European Crohn's and colitis organization (ECCO) guidelines.
3. IBD patients receiving either IFX or ADA.

Exclusion Criteria:

1. Patients missed one-year follow-up or with missed data.
2. Patients having mild IBD according to ECCO guidelines.
3. Patients having any of the Contraindications to the biological Therapy e.g.: latent TB, viral or fungal or bacterial infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Trough concentration of ADA and IFX will be assessed after reaching steady state levels. | 1 month
  Blood Level
myeloid cells 1 (TREM1) levels | 1 month
  predictive biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Principal Investigator — Damanhour University
Locations (1):
- Tropical Medicine department, Ain Shams University Hospitals., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seyedian SS, Nokhostin F, Malamir MD. A review of the diagnosis, prevention, and treatment methods of inflammatory bowel disease. J Med Life. 2019 Apr-Jun;12(2):113-122. doi: 10.25122/jml-2018-0075. PMID 31406511
- [Background] Fluxa, D. and M.T. Abreu, Therapeutic targets in inflammatory bowel disease. Revista Médica Clínica Las Condes, 2019. 30(4): p. 315-322.
- [Background] Shivaji UN, Sharratt CL, Thomas T, Smith SCL, Iacucci M, Moran GW, Ghosh S, Bhala N. Review article: managing the adverse events caused by anti-TNF therapy in inflammatory bowel disease. Aliment Pharmacol Ther. 2019 Mar;49(6):664-680. doi: 10.1111/apt.15097. Epub 2019 Feb 8. PMID 30735257
- [Derived] Kamal ME, Werida RH, Radwan MA, Askar SR, Omran GA, El-Mohamdy MA, Hagag RS. Efficacy and safety of infliximab and adalimumab in inflammatory bowel disease patients. Inflammopharmacology. 2024 Oct;32(5):3259-3269. doi: 10.1007/s10787-024-01508-w. Epub 2024 Jul 10. PMID 38985232